CLINICAL TRIAL: NCT06667050
Title: CAPOX Combined with Sintilimab and Bevacizumab Biosimilar (IBI305) for Neoadjuvant Treatment of Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: a Prospective, Multi-center, Single-arm, Phase II Clinical Trial
Brief Title: CAPOX Plus Sintilimab and Bevacizumab Biosimilar (IBI305) for Neoadjuvant Treatment of Locally Advanced Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, PI, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH241260
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Drug Therapy; sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chemotherapy plus sintilimab and bevacizumab biosimilar (Experimental): capecitabine: 100 mg/m2, Bid, d1-14, q3w; oxaliplatin: 130 mg/m2, iv drip, d1, q3w; sintilimab: 200 mg, iv drip, d1, bevacizumab biosimilar (IBI305) 10mg
  /Kg, iv drip, d1, q3w.
  Interventions: Drug: Chemotherapy plus sintilimab and bevacizumab

INTERVENTIONS:
Drug: Chemotherapy plus sintilimab and bevacizumab — Laparoscopic exploration should be performed to detect occult peritoneal metastases and inspect the primary lesion, liver, diaphragm, pelvic organs, bowel and omentum.
  3 cycles of neoadjuvant therapy will be administered: capecitabine: 100 mg/m2, Bid, d1-14, q3w; oxaliplatin: 130 mg/m2, iv drip, d1, q3w; sintilimab: 200 mg, iv drip, d1, bevacizumab biosimilar (IBI305) 10mg
  /Kg, iv drip, d1, q3w. Radical D2 gastric cancer resection will be performed within 6-8 weeks after the last administration of chemotherapy plus sintilimab and bevacizumab biosimilar (IBI305).
  The adjuvant therapy will start in 4-6 weeks after the surgery, and we recommend adjuvant treatment with CAPOX regimen for up to 3 cycles.

SUMMARY:
Neoadjuvant chemotherapy has been recommended by a series of treatment guidelines for the neoadjuvant treatment of locally advanced G/GEJ cancer. Although with clinical efficacy, the pCR and long-term survival rates are still unsatisfactory and perioperative treatment mode for locally advanced G/GEJ cancer still needs further optimization. In this study, we will explore the efficacy and safety of chemotherapy combined with sintilimab and bevacizumab biosimilar (IBI305) in the neoadjuvant treatment for locally advanced G/GEJ cancer.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, phase II trial. A total of 58 patients will be enrolled. Eligible patients will be registered and receive three cycles of CAPOX plus sintilimab and bevacizumab biosimilar (IBI305) regimen. Radical D2 gastric cancer resection will be performed 6-8 weeks after the last administration of chemotherapy plus plus sintilimab and bevacizumab biosimilar (IBI305). The primary endpoint of the study is the pathological complete response (pCR) rate. Secondary endpoints include R0 resection rate, major pathological response (MPR), event-free survival (EFS), overall survival (OS) and safety profile of the neoadjuvant regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Histologically or cytologically confirmed diagnosis of locally advanced G/GEJ adenocarcinoma (cT3N+/T4aNany M0) as assessed by exploratory laparoscopic surgery, ultrasonography and/or CT/MRI.
3. Resectable G/GEJ cancer, as judged by experienced surgeons.
4. There was no previous antitumor treatment.
5. The expected survival is more than 3 months.
6. ECOG PS≤1.
7. Adequate organ function including the following:

   1. Total bilirubin ≤1.5 times the upper limit of normal (ULN);
   2. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3×ULN;
   3. Alkaline phosphatase≤2.5×ULN (if the tumor invaded the liver, ≤3×ULN);
   4. Serum creatinine≤1.5×ULN;
   5. Serum amylase and lipase≤1.5×ULN;
   6. International standardized ratio (INR)/partial thromboplastin time (PTT)≤1.5×ULN;
   7. Platelet count ≥ 100,000 /mm3;
   8. Hemoglobin (Hb) ≥ 9 g/dL;
   9. Absolute neutrophil count (ANC) ≥ 1500/mm3;
8. Strict contraception.
9. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Undergoing other drug clinical trials or having participated in any drug clinical trials one month before enrollment.
2. Active autoimmune disease or history of refractory autoimmune disease.
3. Receiving corticosteroids (> 10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding the following therapies: steroid hormone replacement therapy (≤10mg/d); local steroid therapy; and short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting.
4. Active or clinically significant cardiac disease:

   1. Congestive heart failure > New York Heart Association (NYHA) class 2;
   2. Active coronary artery disease;
   3. Arrhythmias requiring treatment other than β-blockers or digoxin;
   4. Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment
5. Evidence or history of bleeding diathesis or coagulopathy.
6. Grade 3 bleeding events 4 weeks before enrollment.
7. Thromboembolism or arteriovenous events, such as cerebrovascular events (including transient ischemic attack), deep vein thrombosis or pulmonary embolism, occurred 6 months before enrollment.
8. Currently taking anticoagulants.
9. Gastrointestinal perforation, gastrointestinal obstruction, or uncontrollable diarrhea 6 months before enrollment.
10. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor was cured and no evidence of disease was found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
11. Patients with pheochromocytoma.
12. Patients with a history of HIV infection or active hepatitis B/C.
13. Ongoing > level 2 infection.
14. Symptomatic brain metastasis or meningioma.
15. Unhealed wounds, ulcers or fractures.
16. Renal failure patients requiring blood or peritoneal dialysis.
17. Epileptic that needs medication.
18. Active, symptomatic interstitial pneumonia, pleural or ascites that causes dyspnea (dyspnea ≥ 2 grade).
19. History of organ transplantation (including corneal transplantation).
20. Allergic to research drugs or similar drugs, or suspected allergies.
21. Pregnant or lactating women.
22. Medical, psychological or social conditions can affect the recruitment of patients and evaluation of study results.
23. Other antitumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs. Palliative external irradiation for non-target lesions is allowed.
24. Previously used oxaliplatin, capecitabine, ICIs and anti-angiogenesis drugs;
25. Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery (excluding biliary stents, or percutaneous biliary drainage).
26. Treatment with antitumor Chinese herbal medicine.
27. History of allogeneic blood transfusion within 6 months.
28. Vaccination history within 4 weeks before enrollment.
29. The investigator believes that patients who are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 6 months after the last subject participating in
  defined as the absence of viable tumor cells assessed by histological evaluation criteria after neoadjuvant therapy

SECONDARY OUTCOMES:
R0 resection rate | 6 months after the last subject participating in
  defined as the rate of the complete surgical removal of any residual cancer cells in the tumor bed
MPR rate | 6 months after the last subject participating in
  defined as tumor residual cells ≤10% in the surgical specimen
Event-free survival | 2 years after the last subject participating in
  defined as the time from randomization to occurrence of a major adverse clinical event, such as failure to achieve remission, relapse, and death during remission.
Overall survival | 2 years after the last subject participating in
  defined as the time from randomization to occurrence of death during remission.
Treatment-related adverse events | 3 months after the last administration of drugs
  Treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No